CLINICAL TRIAL: NCT06850090
Title: Neoadjuvant Radiotherapy for Rectal Adenocarcinoma With Capecitabine Versus TAS-102 (Neo-REACT): A Multi-center, Randomized, Phase III Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Radiation Oncology Department, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-026-02
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer; Rectal Cancer Patients
MeSH Terms: conditions — Rectal Neoplasms | interventions — trifluridine tipiracil drug combination; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TAS-102 group (Experimental): Neoadjuvant long-course radiotherapy combined with TAS-102
  Interventions: Combination Product: TAS-102
- Capecitabine group (Active Comparator): Neoadjuvant long-course radiotherapy combined with capecitabine
  Interventions: Combination Product: Capecitabine

INTERVENTIONS:
Combination Product: TAS-102 — Radiotherapy:
  1. Radiotherapy Technique: Three-dimensional conformal radiotherapy (3D-CRT), intensity-modulated radiotherapy (IMRT), or volume modulated arc therapy (VMAT);
  2. Radiotherapy Dose and Fractionation Schedule: Conventional fractionation with external beam irradiation at a dose of 50 Gy delivered in 25 fractions over 5 weeks.
  Synchronous Chemotherapy:
  Concurrent administration of TAS-102 at a dose of 35 mg/m² twice daily at the 1st, 3rd and 5th week of radiotherapy.
  Intermittent Consolidation Chemotherapy:
  Oxaliplatin at 85 mg/m² on day 1 combined with TAS-102 at 35 mg/m² twice daily from day 1 to day 5, repeated every 14 days for a total of 6 cycles.
  Surgery:
  The operation follows the principle of TME. The type of surgery depends on the location and extent of the primary tumor.
  Postoperative adjuvant therapy:
  Two cycles of CapeOX (Oxaliplatin 130 mg/m2 on day 1+ capecitabine 1000 mg/m2 twice a day on days 1-14, q3w).
  Arms: TAS-102 group
Combination Product: Capecitabine — Radiotherapy:
  1. Radiotherapy Technique: Three-dimensional conformal radiotherapy (3D-CRT), intensity-modulated radiotherapy (IMRT), or volume modulated arc therapy (VMAT);
  2. Radiotherapy Dose and Fractionation Schedule: Conventional fractionation with external beam irradiation at a dose of 50 Gy delivered in 25 fractions over 5 weeks.
  Synchronous Chemotherapy:
  Capecitabine administered orally at a dose of 825 mg/m² twice daily on days of radiotherapy.
  Intermittent Consolidation Chemotherapy:
  Oxaliplatin at 130 mg/m² on day 1 combined with capecitabine at 1000 mg/m² twice daily from day 1 to day 14, repeated every 21 days for a total of 4 cycles.
  Surgery:
  The operation follows the principle of TME. The type of surgery depends on the location and extent of the primary tumor.
  Postoperative adjuvant therapy: Two cycles of CapeOX (Oxaliplatin 130 mg/m2 on day 1+ capecitabine 1000 mg/m2 twice a day on days 1-14, q3w)
  Arms: Capecitabine group

SUMMARY:
Neoadjuvant fluoropyrimidine-based chemoradiotherapy followed by total mesorectal excision (TME) is the standard of care for locally advanced rectal cancer (LARC); however, pathologic complete response (pCR) rates are low. Trifluridine/tipiracil (TAS-102) is a new oral anti-tumor oral formulation of nucleoside analogue, trifluridine (FTD), and a thymidine phosphorylase inhibitor, tipiracil (TPI). Previous studies have shown that TAS-102 has shown clinically relevant activity after fluoropyrimidine failure in colorectal cancer and may thus be of increased efficacy compared with current standard capecitabine chemoradiation. Also, a phase 2 trials conducted by our team have demonstrated that neoaduvant TAS-102 concurrent with long-course radiotherapy could lead to a high pCR rate of 32% with acceptable toxicity for LARC patients. Herein, we will conduct this multicenter, randomized controlled, phase III trial to explore the safety and efficacy benefit of TAS-102 concurrent with long-course radiotherapy for LARC.

DETAILED DESCRIPTION:
Neoadjuvant fluoropyrimidine-based chemoradiotherapy (nCRT) followed by TME is the standard care for LARC. However, the tumor responses to nCRT cover a wide spectrum and the complete pathologic response rate varies from 8% to 20%. The low rate of pCR after neoadjuvant therapy could not satisfy patients with distal rectal cancer who want to keep anal function. Therefore, currently, the addition of other agents to 5-FU or capecitabine as components of the multimodality treatment for LARC outside of clinical trials is not recommended in clinical practice. TAS-102 is a new oral anti-tumor oral formulation of nucleoside analogue, FTD, and a thymidine phosphorylase inhibitor, TPI. TPI improves the bioavailability and ensures sufficient blood concentrations of FDT. Previous studies have shown that TAS-102 has shown clinically relevant activity after fluoropyrimidine failure in colorectal cancer and may thus be of increased efficacy compared with current standard capecitabine chemoradiation. Also, a phase 2 trials conducted by our team have demonstrated that neoaduvant TAS-102 concurrent with long-course radiotherapy could lead to a high pCR rate of 32% with acceptable toxicity for LARC patients. Herein, we will conduct this multicenter, randomized controlled, phase III trial to explore the safety and efficacy benefit of TAS-102 concurrent with long-course radiotherapy for LARC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 75 years of either sex.
2. Histologically confirmed rectal adenocarcinoma with the following conditions:

   1. Clinical stage II (T3-4, N-) or III (any T, N+) as determined by MRI.
   2. The tumor is located within 12 cm from the anal margin, with at least one high-risk factors (ie, extramural vascular invasion [EMVI+], mesorectal fascia involved [MRF+], cT4, cN2, lateral lymph nodes, tumor deposit, or tumor located in the lower rectum [≤5 cm from the anal verge]).
3. No other types of rectal cancer (e.g., sarcoma, lymphoma, carcinoid, squamous cell carcinoma) or synchronous colon cancer.
4. Presence of measurable lesions that meet RECIST v1.1 criteria for evaluation.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
6. Estimated life expectancy > 6 months.

Exclusion Criteria:

1. Patients of dMMR or MSI-H status.
2. Unexplained myelosuppression.
3. Evidence of distant metastasis and inguinal lymph node metastasis based on comprehensive chest and abdominal CT or whole-body PET-CT scans. Retroperitoneal lymph nodes above the iliac vessel bifurcation are considered distant metastasis.
4. Active autoimmune disease or history of autoimmune disease.
5. Uncontrolled cardiac symptoms or diseases.
6. History of other malignancies, except for cured basal cell carcinoma of the skin and cervical carcinoma in situ.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 1 year
  The primary outcomes is CR rate, which is the sum of the number of patients with a pCR who undergo surgery plus the number of patients with a cCR who undergo watch-and-wait divided by the total number of evaluable patients.

SECONDARY OUTCOMES:
The incidence of 3-4 grade adverse reactions | 1 year
  The adverse reactions are graded and recorded according to the National Cancer Institute General Terminology for Adverse Events (CTCAE) Version 5.0.
3-year recurrence-free survival (RFS) | 3 year
  3-year RFS is measured from randomization to the first occurrence of recurrence or last follow-up.
3-year overall survival (OS) | 3 year
  3-year OS is measured from randomization to death due to any cause or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Docter, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No